CLINICAL TRIAL: NCT05076071
Title: Clinical Value of Next Generation Sequencing in Chinese Childhood Solid Tumors: A Multicenter Study
Brief Title: Clinical Value of Next Generation Sequencing in Chinese Childhood Solid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yizhuo Zhang (Other)
Responsible Party: Sponsor-Investigator, Yizhuo Zhang, proffesor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: SunYat-sen U
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Pediatric, Solid Tumors, NGS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: NGS — Next Generation Sequencing

SUMMARY:
Samples of 200 patients with pediatric malignant solid tumors will prospectively be collected. Selected samples are sufficient for next generation sequencing(NGS) and available for follow-up information. Multi-omics techniques such as DNA and RNA panel will be used to study driver genes for the development of malignant solid tumors in children, and to explore the pathogenic mechanism. The aim of this study is to explore new biomarkers for the diagnosis and treatment for childhood malignant solid tumors.

DETAILED DESCRIPTION:
DNA and RNA extracted from tumor tissues and leukocytes will be analyzed by Onco PanScan/whole exon sequencing(Genetronhealth), and comprehensive gene mutation information such as single nucleotide variation, insertion deletion mutation, gene copy number variants and structure variants will be obtained.

Through in-depth mining of genomic data generated by clinical tumor tissue detection, the differences among different subtypes of pediatric solid tumors in TCGA data will be compared with previous studies. Combined with clinical pathological and molecular subtyping results, auxiliary diagnosis was performed. Analyzing therapeutic targets and identifying pathogenic cancer-predisposing variants may provide molecular reference for children's malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are diagnosed by histology and pathology as pediatric malignant solid tumors (including soft tissue sarcoma, osteosarcoma, pediatric glioma, neuroblastoma, nephroblastoma, retinoblastoma, hepatoblastoma, atypical teratoid/rhabdomymoma, embryonal tumor, etc.);
2. Age: < 18 years old;
3. Eastern Cooperative Oncology Group (ECOG) PS score: 0-2, estimated survival >6 months;
4. Complete clinical laboratory examination and pathological examination information of patients;
5. Patients can be evaluated on time, and samples can be obtained throughout the whole test process;
6. Informed consent signed by the patient or his/her legal representative shall be obtained after the patient is informed of the project;

Exclusion Criteria:

1. As determined by the investigator, the patient had other major diseases that might affect follow-up and short-term survival;
2. Any social/psychological problems that the researcher determines are not suitable for the study;

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 200
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-07-06 (Estimated); Study Completion 2023-08-06 (Estimated)

PRIMARY OUTCOMES:
Mutation characteristics of malignant solid tumors in Chinese children. | 2021.8-2023.8

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu S, Zhang Y, Zhang W, Huang J, Yang C, Wang J, Gao J, Guo X, Yuan X, Chen S, Sun F, Cheng H, Yao W, Dong K, Guo H, Sun X, Li H, Chen K, Lan H, Zhen Z, Zhu J, Zhang X, Que Y, Yan S, Ma J, Li J, Zhu D, Wang H, Wang S, Zhang Y. Precision Medicine Program in Chinese Pediatric Patients With Sarcoma. JCO Precis Oncol. 2026 Jan;10:e2500428. doi: 10.1200/PO-25-00428. Epub 2026 Jan 14. PMID 41533994